CLINICAL TRIAL: NCT05516810
Title: The Accuracy of Ultrasound Diagnosis of Hydatidiform Moles
Status: Active, not recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 136133
Record Dates: First submitted 2022-07-27; First posted 2022-08-26 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hydatidiform Mole (Diagnosis); Abortion, Spontaneous; Missed Abortion; Incomplete Miscarriage; Miscarriage in First Trimester
Keywords: ultrasonography; pregnancy, first trimester; molar; miscarriage; hydatidiform
MeSH Terms: conditions — Hydatidiform Mole; Disease; Abortion, Spontaneous; Abortion, Missed; Abortion, Incomplete

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study assessing which ultrasound findings are best at excluding a molar pregnancy in first trimester miscarriage.

DETAILED DESCRIPTION:
The objectives of this study are to establish the accuracy of ultrasound for the diagnosis of HMs, assess prevalence of these ultrasound features in early pregnancy failure (missed-miscarriages and incomplete miscarriages), and establish which ultrasound signs are the best predictor of HMs on histopathology. The findings of this study will allow us to improve the early diagnosis of HMs by ultrasound therefore allowing us to tailor our counselling and clinical management.

All women attending the EPUs and with findings of an early embryonic demise or incomplete miscarriage on transvaginal scan (either by dates or by scan findings) will be eligible to take part in the study. The NICE criteria to diagnose miscarriage will be used.

Diagnostic criteria derived from retrospective studies will be used to make the diagnosis of suspected HMs on ultrasound and the presence or absence of these features specifically noted. All participants will be scanned by specialist Gynaecologists who are members of the research team, or the direct clinical care team.

Women with suspected HMs on ultrasound will be advised to undergo surgical management of miscarriage, which is in line with current national clinical guidance and maximises the chance of histological diagnosis. All other participants will be offered surgical, medical or expectant management as per standard clinical practice. All women who opt for surgical management, or in whom any pregnancy tissue is available, will have their pregnancy tissue sent for histology, as per national guidance. We will then compare the ultrasound findings with the final histological diagnosis for those women with histopathology specimens and will phone those participants without histopathology specimens to check that their pregnancy tests have reverted to negative 3 weeks after their miscarriage so as to exclude persistent GTN as per standard clinical practice. In addition to this we will perform a blood test for checking pregnancy hormones, beta HCG to assess the correlation between these levels and histologically diagnosed hydatiform moles.

All eligible women will be invited to participate in the study and be provided with written consent to have their clinical data included in the study following their ultrasound scan.

Participation in the study will be voluntary and refusal to participate will not affect patients' care. Furthermore, taking part in the study will involve an additional blood test, but no other additional interventions over their routine clinical care; however, it will include personal data collection for the purpose of the study. All identifiable data will be anonymised.

ELIGIBILITY:
Inclusion Criteria:

* less than 16 weeks gestation by last menstrual period or by ultrasound
* singleton pregnancy
* ultrasound diagnosis of early embryonic demise or incomplete miscarriage or suspected molar pregnancy.

Exclusion Criteria:

* Women declining participation and follow up
* Women who refuse transvaginal scan
* Multiple pregnancy
* Ectopic pregnancy
* Pregnancy of unknown location
* Those unable to understand English to an adequate degree to understand and consent to participation in this study

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women diagnosed with embryonic demise, incomplete miscarriage or suspected molar pregnancy within two UK hospitals' early pregnancy units
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
histological diagnosis of molar pregnancy yes / no | within a month post miscarriage
  binary outcome measure
hCG undetectable in the urine yes / no | up to 2 months post miscarriage
  Negative pregnancy test post miscarriage for those with no tissue available for histology

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Ross, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - University College London Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No
no plan to share participant data with other researchers